CLINICAL TRIAL: NCT02083315
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Explore the Pharmacokinetics and Pharmacodynamics of TRV130, Morphine, and Placebo in Healthy Adult Male Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics of TRV130, Morphine, and Placebo in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP130-1003
Record Dates: First submitted 2014-02-24; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Pain, Acute
Keywords: acute pain, analgesia, respiratory drive, ventilator response to hypercapnia, pupillometry
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- TRV130 1.5 mg (Experimental): TRV130 1.5 mg IV x 1 dose
  Interventions: Drug: TRV130 1.5 mg
- TRV130 3 mg (Experimental): TRV130 3 mg IV x 1 dose
  Interventions: Drug: TRV130 3 mg
- TRV130 4.5 mg (Experimental): TRV130 4.5 mg IV x 1 dose
  Interventions: Drug: TRV130 4.5 mg
- Morphine (Active Comparator): Morphine 10 mg IV x 1 dose
  Interventions: Drug: Morphine 10 mg
- Placebo (Placebo Comparator): Dextrose 5% in water IV x 1 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRV130 1.5 mg — TRV130 1.5 mg IV x 1 dose
  Arms: TRV130 1.5 mg
Drug: TRV130 3 mg — TRV130 3 mg IV x 1 dose
  Arms: TRV130 3 mg
Drug: TRV130 4.5 mg — TRV130 4.5 mg IV x 1 dose
  Arms: TRV130 4.5 mg
Drug: Morphine 10 mg — Morphine 10 mg IV x 1 dose
  Arms: Morphine
Drug: Placebo — Dextrose 5% in water IV x 1 dose
  Arms: Placebo

SUMMARY:
This study is designed to compare TRV130 to placebo and morphine to learn about its effects on pain relief and side effects.

DETAILED DESCRIPTION:
This study will explore the pharmacokinetics, pharmacodynamics (PD), safety and tolerability of TRV130.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Healthy adult males age 18 - 50 years, BMI 19-32 kg/m2
* Acceptable duration of cold pain test results at screening

Exclusion Criteria:

* Clinically significant medical illness or physical exam findings
* Active dermatological conditions or skin trauma on the non-dominant hand, or peripheral vascular disease
* Partial blindness, keratoconus, nystagmus or any other ophthalmic condition which could interfere with pupillometry
* Use of tobacco or nicotine within 6 months prior to screening
* History of recent (within 6 months) drug or alcohol abuse, as defined in DSM-IV-TR

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cold Pain Test | 8 hours postdose

SECONDARY OUTCOMES:
Ventilatory Response to Hypercapnia | 4 hours postdose
Pupillometry | 8 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: David G Soergel, MD, Study Chair — Trevena Inc.
Locations (1):
- CRI Lifetree, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Soergel DG, Subach RA, Burnham N, Lark MW, James IE, Sadler BM, Skobieranda F, Violin JD, Webster LR. Biased agonism of the mu-opioid receptor by TRV130 increases analgesia and reduces on-target adverse effects versus morphine: A randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Pain. 2014 Sep;155(9):1829-1835. doi: 10.1016/j.pain.2014.06.011. Epub 2014 Jun 19. PMID 24954166